CLINICAL TRIAL: NCT02233322
Title: Iron Therapy for Autosomal Dominant Hypophosphatemic Rickets: A Pilot
Brief Title: Iron Therapy for Autosomal Dominant Hypophosphatemic Rickets: A Pilot Project.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Michael Econs, Professor of Endocrinology and Metabolism, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRON/ADHR
Record Dates: First submitted 2014-08-27; First posted 2014-09-08 (Estimated); Last update posted 2019-11-14 (Actual); Status verified 2019-11

CONDITIONS: Autosomal Dominant Hypophosphatemic Rickets
Keywords: ADHR; Rickets; Hypophosphatemia
MeSH Terms: conditions — Hypophosphatemic Rickets, Autosomal Dominant; Rickets; Hypophosphatemia | interventions — Iron; ferrous sulfate; ferrous gluconate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- iron supplements (Experimental): all subjects will receive iron supplementation based on iron levels in blood
  Interventions: Dietary Supplement: Iron

INTERVENTIONS:
Dietary Supplement: Iron — All subjects will receive iron supplementation based on iron levels in the blood
  Other Names: Ferrous Sulfate; Ferrous Gluconate

SUMMARY:
The purpose of the study is to gain a better understanding of the effect of iron on fibroblast growth factor 23 (FGF23) in the inherited disorder, autosomal dominant hypophosphatemic rickets (ADHR). ADHR is an inherited disorder in which the body makes too much FGF 23 and causes low blood phosphorus levels and bone problems such as rickets (bowed legs in children) or bone pain and weakness in adults. This study is to test whether or not giving iron helps correct the high FGF23 and there by correcting the phosphate problem.

DETAILED DESCRIPTION:
Iron will be provided in an open label treatment to all enrolled subjects. Iron levels will be monitored in blood and doses adjusted with the target of getting the iron levels to or a little above 100 mcg/dl.

The study will look to see if there is a decrease of FGF23 level. It will also look at how long does it take to decrease the level of FGF 23 and how long it takes for the serum and urine phosphate to normalize.

ELIGIBILITY:
Inclusion Criteria:

* FGF Mutation in either Arginine 176 or arginine 179
* able and willing to provide consent or have a parent that is able/willing to consent, if a minor
* either serum iron <50mcg/dl (regardless of phosphate or intact FGF23 concentration); or iron between 500 and 100mcg/dl with serum phosphorus value below 3.0mg/dl for adults or less than or equal to 0.5 mg/dl the lower limit of normal for age in children and intact FGF23 about 30pg/ml
* age >2 years
* May be receiving treatment with phosphate and calcitriol, but must be willing to undergo dose adjustments by the investigators if iron resolves the phosphate wasting defect.

Exclusion Criteria:

* malignancy within the last 5 years, except treated squamous or basal cell skin carcinoma
* terminal illness/hospice.
* severe end-organ disease, e.g. cardiovascular, pulmonary, etc, which may limit ability to complete study.

estimated GFR <45ml/min/1.73m2, calculated using MDRD formula for adults or modified Schwartz equation for children

* pregnancy or plan on becoming pregnant

Min Age: 25 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2014-08; Primary Completion 2019-11-12 (Actual); Study Completion 2019-11-12 (Actual)

PRIMARY OUTCOMES:
Does increasing serum iron concentrations above 100 mcg/dl in patients with ADHR result in a decrease in intact FGF23. | FGF23 will be measured at 1, 2, 3, 6, 9, and 12 months
  Perform a pilot study in ADHR patients with low serum iron concentrations (defined below) to determine if increasing serum iron concentrations above 100 mcg/dl results in a decrease in intact FGF23 (primary endpoint) and C-terminal FGF23 concentrations by at least 20% and normalizes serum phosphorus and TMP/GFR (tubular maximum phosphate reabsorption/ glomerular filtration rate) within 6 months of attaining goal iron concentrations.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Econs, M.D., Principal Investigator — Indiana University School of Medicine
Locations (1):
- Indiana University School of Medicine, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] White KE, Carn G, Lorenz-Depiereux B, Benet-Pages A, Strom TM, Econs MJ. Autosomal-dominant hypophosphatemic rickets (ADHR) mutations stabilize FGF-23. Kidney Int. 2001 Dec;60(6):2079-86. doi: 10.1046/j.1523-1755.2001.00064.x. PMID 11737582
- [Background] Imel EA, Hui SL, Econs MJ. FGF23 concentrations vary with disease status in autosomal dominant hypophosphatemic rickets. J Bone Miner Res. 2007 Apr;22(4):520-6. doi: 10.1359/jbmr.070107. PMID 17227222
- [Background] Imel EA, Peacock M, Gray AK, Padgett LR, Hui SL, Econs MJ. Iron modifies plasma FGF23 differently in autosomal dominant hypophosphatemic rickets and healthy humans. J Clin Endocrinol Metab. 2011 Nov;96(11):3541-9. doi: 10.1210/jc.2011-1239. Epub 2011 Aug 31. PMID 21880793
- [Background] Farrow EG, Yu X, Summers LJ, Davis SI, Fleet JC, Allen MR, Robling AG, Stayrook KR, Jideonwo V, Magers MJ, Garringer HJ, Vidal R, Chan RJ, Goodwin CB, Hui SL, Peacock M, White KE. Iron deficiency drives an autosomal dominant hypophosphatemic rickets (ADHR) phenotype in fibroblast growth factor-23 (Fgf23) knock-in mice. Proc Natl Acad Sci U S A. 2011 Nov 15;108(46):E1146-55. doi: 10.1073/pnas.1110905108. Epub 2011 Oct 17. PMID 22006328
- [Background] Econs MJ, McEnery PT. Autosomal dominant hypophosphatemic rickets/osteomalacia: clinical characterization of a novel renal phosphate-wasting disorder. J Clin Endocrinol Metab. 1997 Feb;82(2):674-81. doi: 10.1210/jcem.82.2.3765. PMID 9024275
- [Background] Schouten BJ, Doogue MP, Soule SG, Hunt PJ. Iron polymaltose-induced FGF23 elevation complicated by hypophosphataemic osteomalacia. Ann Clin Biochem. 2009 Mar;46(Pt 2):167-9. doi: 10.1258/acb.2008.008151. Epub 2009 Jan 16. PMID 19151167
- [Background] Schouten BJ, Hunt PJ, Livesey JH, Frampton CM, Soule SG. FGF23 elevation and hypophosphatemia after intravenous iron polymaltose: a prospective study. J Clin Endocrinol Metab. 2009 Jul;94(7):2332-7. doi: 10.1210/jc.2008-2396. Epub 2009 Apr 14. PMID 19366850
- [Background] Shimizu Y, Tada Y, Yamauchi M, Okamoto T, Suzuki H, Ito N, Fukumoto S, Sugimoto T, Fujita T. Hypophosphatemia induced by intravenous administration of saccharated ferric oxide: another form of FGF23-related hypophosphatemia. Bone. 2009 Oct;45(4):814-6. doi: 10.1016/j.bone.2009.06.017. Epub 2009 Jun 23. PMID 19555782
- [Background] Bianchine JW, Stambler AA, Harrison HE. Familial hypophosphatemic rickets showing autosomal dominant inheritance. Birth Defects Orig Artic Ser. 1971 May;7(6):287-95. No abstract available. PMID 5173181
- [Background] Econs MJ, McEnery PT, Lennon F, Speer MC. Autosomal dominant hypophosphatemic rickets is linked to chromosome 12p13. J Clin Invest. 1997 Dec 1;100(11):2653-7. doi: 10.1172/JCI119809. PMID 9389727
- [Background] Schwartz GJ, Munoz A, Schneider MF, Mak RH, Kaskel F, Warady BA, Furth SL. New equations to estimate GFR in children with CKD. J Am Soc Nephrol. 2009 Mar;20(3):629-37. doi: 10.1681/ASN.2008030287. Epub 2009 Jan 21. PMID 19158356
- [Background] Walton RJ, Bijvoet OL. Nomogram for derivation of renal threshold phosphate concentration. Lancet. 1975 Aug 16;2(7929):309-10. doi: 10.1016/s0140-6736(75)92736-1. No abstract available. PMID 50513
- [Background] Ichikawa S, Imel EA, Kreiter ML, Yu X, Mackenzie DS, Sorenson AH, Goetz R, Mohammadi M, White KE, Econs MJ. A homozygous missense mutation in human KLOTHO causes severe tumoral calcinosis. J Clin Invest. 2007 Sep;117(9):2684-91. doi: 10.1172/JCI31330. PMID 17710231
- [Background] Imel EA, DiMeglio LA, Hui SL, Carpenter TO, Econs MJ. Treatment of X-linked hypophosphatemia with calcitriol and phosphate increases circulating fibroblast growth factor 23 concentrations. J Clin Endocrinol Metab. 2010 Apr;95(4):1846-50. doi: 10.1210/jc.2009-1671. Epub 2010 Feb 15. PMID 20157195
- [Background] Imel EA, Peacock M, Pitukcheewanont P, Heller HJ, Ward LM, Shulman D, Kassem M, Rackoff P, Zimering M, Dalkin A, Drobny E, Colussi G, Shaker JL, Hoogendoorn EH, Hui SL, Econs MJ. Sensitivity of fibroblast growth factor 23 measurements in tumor-induced osteomalacia. J Clin Endocrinol Metab. 2006 Jun;91(6):2055-61. doi: 10.1210/jc.2005-2105. Epub 2006 Mar 21. PMID 16551733
- [Background] Sabbagh, Y., Tenenhouse HS, Econs, MJ, Mendelian Hypophosphatemias, in The Metabolic and Molecular Basis of Inherited Disease, C.R.S.e. al, Editor. 2008, McGraw-Hill: New York.
- [Background] White, K.E. and M.J. Econs, Fibroblast growth factor-23 (FGF23), in Primer on the Metabolic Bone Diseases and Disorders of Mineral Metabolism. 2013, Wiley-Blackwell. p. 188-194.
- [Background] ADHR Consortium. Autosomal dominant hypophosphataemic rickets is associated with mutations in FGF23. Nat Genet. 2000 Nov;26(3):345-8. doi: 10.1038/81664. PMID 11062477
- [Derived] Imel EA, Liu Z, Coffman M, Acton D, Mehta R, Econs MJ. Oral Iron Replacement Normalizes Fibroblast Growth Factor 23 in Iron-Deficient Patients With Autosomal Dominant Hypophosphatemic Rickets. J Bone Miner Res. 2020 Feb;35(2):231-238. doi: 10.1002/jbmr.3878. Epub 2019 Oct 25. PMID 31652009